CLINICAL TRIAL: NCT00150748
Title: An Open-label, Multicenter, Follow-up Study to Evaluate the Safety and Efficacy of Levetiracetam (LEV) (Oral Tablets of 166, 250 or 500 mg b.i.d.), at Individualized Doses up to a Maximum of 4000 mg/Day (or 80 mg/kg/Day for Children and Adolescents Less Than 50 kg), in Children (≥ 4 Years Old), Adolescents and Adults Suffering From Primary Generalized Seizures
Brief Title: Long Term Follow up Treatment With Levetiracetam in Subjects of 4 Years and Older With Generalized Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N167; 2004-001997-13 (EudraCT Number)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Generalized Epilepsy
Keywords: Generalized Epilepsy, Primary Generalized Seizures; Keppra, Levetiracetam
MeSH Terms: conditions — Epilepsy, Generalized | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental): Subjects received treatment up to 1764 days during the Evaluation Period. Up to 4000 mg/day (or 80 mg/kg/day for children and adolescents less than 50 kg). Oral tablets of 166, 250, or 500 mg Levetiracetam twice daily (b.i.d.).
  Interventions: Drug: Levetiracetam 166 mg; Drug: Levetiracetam 250 mg; Drug: Levetiracetam 500 mg

INTERVENTIONS:
Drug: Levetiracetam 166 mg — * Active Substance: Levetiracetam
  * Pharmaceutical Form: Tablet
  * Concentration: 166 mg
  * Route of Administration: Oral use
Drug: Levetiracetam 250 mg — * Active Substance: Levetiracetam
  * Pharmaceutical Form: Tablet
  * Concentration: 250 mg
  * Route of Administration: Oral use
Drug: Levetiracetam 500 mg — * Active Substance: Levetiracetam
  * Pharmaceutical Form: Tablet
  * Concentration: 500 mg
  * Route of Administration: Oral use

SUMMARY:
An open-label, follow-up study to evaluate the safety and efficacy of levetiracetam (LEV), in children (≥ 4 years old), adolescents and adults suffering from primary generalized seizures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children, adolescents and adults having completed the final visit of a previous study with levetiracetam (LEV)
* Subjects who were/are suffering from primary generalized (type II) epileptic seizures
* Subjects for whom the Investigator believes a reasonable benefit (efficacy or tolerability) from the long-term administration of LEV may be expected

Exclusion Criteria:

* Known clinically significant acute or chronic illness, for example: cardiac, renal or hepatic dysfunction, etc., which may impair reliable participation in the trial or necessitate the use of medication not allowed by protocol
* Concomitant use of any drug with possible central nervous system effects unless at a stable dose
* Concomitant use of any drug (other than hormonal treatment and the subject's normal anti-epileptic drugs (AEDs) that may influence the metabolism of the concomitant AED(s), except if the dose has been stable before entry in the study for sufficient length of time

Ages: 4 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 217 (Actual)
Dates: Start 2001-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects having at least 6 months of seizure freedom at any time during the Evaluation Period | Evaluation Period
Percentage of subjects having at least 6 months of seizure freedom at any time during the Evaluation Period | Evaluation Period

SECONDARY OUTCOMES:
Number of subjects remaining seizure-free, for the All intent-to-treat (ITT) population, and Tonic-Clonic, Myoclonic, and Absence subpopulations since the beginning of this study N167 (Visit 1) during the Evaluation Period | From Visit 1 to the end of the Evaluation Period
Percentage of subjects remaining seizure-free, for the All intent-to-treat (ITT) population, and Tonic-Clonic, Myoclonic, and Absence subpopulations since the beginning of this study N167 (Visit 1) during the Evaluation Period | From Visit 1 to the end of the Evaluation Period
Reduction from N01057 or N166 Baseline to the Evaluation Period in seizure frequency per week for Tonic-Clonic subpopulation seizures types | From N01057 or N166 Baseline to the Evaluation Period
Percentage reduction from N01057 or N166 Baseline to the Evaluation Period in seizure frequency per week for Tonic-Clonic subpopulation seizures types | From N01057 or N166 Baseline to the Evaluation Period
Reduction from N01057 or N166 Baseline to the Evaluation Period in seizure days per week for the ITT population, and Absence and Myoclonic subpopulations | From N01057 or N166 Baseline to the Evaluation Period
Percentage reduction from N01057 or N166 Baseline to the Evaluation Period in seizure days per week for the ITT population, and Absence and Myoclonic subpopulations | From N01057 or N166 Baseline to the Evaluation Period
Categorical percentage reduction from Baseline to the Evaluation Period in seizure days per week for the ITT population, and Absence and Myoclonic subpopulations | Evaluation Period
Categorical percentage reduction from Baseline to the Evaluation Period in seizure frequency per week for Tonic-Clonic subpopulation seizures types | Evaluation Period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877-822-9493

REFERENCES:
- [Derived] Delanty N, Jones J, Tonner F. Adjunctive levetiracetam in children, adolescents, and adults with primary generalized seizures: open-label, noncomparative, multicenter, long-term follow-up study. Epilepsia. 2012 Jan;53(1):111-9. doi: 10.1111/j.1528-1167.2011.03300.x. Epub 2011 Nov 2. PMID 22050371